CLINICAL TRIAL: NCT07127289
Title: A Prospective, Single-Arm, Single-Center Study of Autologous Hematopoietic Stem Cell Infusion for Prolonged Cytopenia After CAR-T Cell Therapy
Brief Title: Autologous Hematopoietic Stem Cell Infusion for Prolonged Cytopenia After CAR-T Cell Therapy
Acronym: ICAHT-001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025001
Record Dates: First submitted 2025-07-30; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Prolonged Cytopenia Following CAR-T Therapy
Keywords: Stem cell; CAR-T; prolonged cytopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous hematopoietic stem cell infusion (Experimental)
  Interventions: Biological: Autologous hematopoietic stem cell infusion

INTERVENTIONS:
Biological: Autologous hematopoietic stem cell infusion — Autologous hematopoietic stem cell infusion (0.5-3.0×10^6/kg)

SUMMARY:
This is a prospective, single-arm, single-center clinical study designed to evaluate the safety of autologous hematopoietic stem cell infusion for the treatment of prolonged cytopenia following CAR-T cell therapy. Approximately 20 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent form (ICF).
2. Age ≥ 18 years.
3. Diagnosis of multiple myeloma according to the International Myeloma Working Group (IMWG) criteria.
4. Prior treatment with CAR-T cell therapy and currently in remission or, in the opinion of the investigator, with refractory/progressive disease not requiring salvage therapy.
5. Presence of grade 3-4 cytopenia (absolute neutrophil count < 1.0 × 10⁹/L, or platelet count < 50 × 10⁹/L, or hemoglobin < 80 g/L) either persisting or newly developed between day 30 and day 90 after CAR-T cell infusion; or deemed suitable for inclusion by the investigator based on clinical judgment.
6. Availability of ≥ 1 × 10⁶/kg autologous hematopoietic stem cells in reserve.

Exclusion Criteria:

1. Known intolerance, hypersensitivity, or contraindication to autologous hematopoietic stem cell infusion.
2. Active hepatitis B or hepatitis C virus infection.
3. Known HIV infection.
4. Life expectancy <6 months.
5. Woman who are pregnant or breastfeeding.
6. Evidence of uncontrolled dysfunction of heart, lung, brain, and other important organs.
7. Any other conditions that are not eligible for the trial in the judgement of the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Changes in Neutrophil Counts After Autologous Stem Cell Infusion | up to 6 months after infusion
  Evaluate changes in neutrophil counts following autologous hematopoietic stem cell infusion.
Changes in Platelet Counts After Autologous Stem Cell Infusion | up to 6 months after infusion
  Evaluate changes in platelet counts following autologous hematopoietic stem cell infusion.
Changes in Hemoglobin Levels After Autologous Stem Cell Infusion | up to 6 months after infusion
  Evaluate changes in hemoglobin levels following autologous hematopoietic stem cell infusion.
Incidence and Severity of Adverse Events Following Autologous Stem Cell Infusion | up to 6 months after infusion
  Assess safety by monitoring infusion-related adverse events, graded according to CTCAE v5.0.

SECONDARY OUTCOMES:
Incidence of Infections After Autologous Stem Cell Infusion | up to 6 months after infusion
  Evaluate the frequency and types of infections following stem cell infusion, including bacterial, viral, and fungal infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No